Investigation of the feasibility of an articulated laparoscopic camera system - Precision Robotics' Sirius Robotic Flexible Endoscopic System in gynaecological laparoscopic surgery

NCT ID not yet assigned Unique Protocol ID: PRHK HKU-GHK IRB 2021-01 Dated 18 February, 2021



# Study on Precision Robotics' Sirius Robotic Flexible Endoscopic System in Gynaecological Laparoscopic Surgery

## **Information Sheet and Consent**

### What is the Sirius Robotic Flexible Endoscopic System?

- Precision Robotics' Sirius Robotic Flexible Endoscopic System is a fully integrated compact 3D laparoscopic camera system with a flexible robotic tip that can change its viewing direction.
- The articulated tip has three degrees of freedom enabling C and S-shaped bending providing a wider field of view compared to conventional laparoscopes.
- This flexibility and wider field of view can potentially help gynaecological laparoscopic surgeons perform their surgery better, especially for advanced laparoscopic procedures such as Single Incision Laparoscopic Surgery(SILS) and Vaginal Natural Orifice Transluminal Surgery(vNOTEs).
- The Sirius Robotic Flexible Endoscopic System has completed all preclinical testing as well as safety checks.
- Clinical trials are in progress and GHK has been selected as one of the centres for clinical trials in Hong Kong.

#### Aim of the Study

- To assess the safety, reliability and efficacy of an articulated laparoscopic camera system Precision Robotics' Sirius Robotic Flexible Endoscopic System in gynaecological laparoscopic surgery particularly for Single Incision Laparoscopic Surgery(SILS) and Vaginal Natural Orifice Transluminal Endoscopy(vNOTEs).
- The aim of this clinical trial is to assess if the Sirius Robotic Flexible Endoscopic System can replace the conventional endoscope in gynaecological laparoscopic procedures.
- The only difference in the laparoscopic procedure is the replacement of the conventional endoscope by the Sirius Robotic Flexible Endoscopic System. All other instruments and procedures remain the same.

### Participation in the trial

- As you are about to undergo a laparoscopic gynaecological procedure, you have been invited to participate in the trial.
- Photographic and/or video images may be taken during the operation for education/ research/ documentation purpose. Your name and ID number will not be recorded and so your identity will not be disclosed. Please inform the staff if you have any objection.
- Participation in the trial is voluntary, and your laparoscopic surgery will be done in the usual manner with a conventional endoscope should you choose not to participate in the trial.



• The Sirius Robotic Flexible Endoscopic System will be used during the laparoscopic procedure, and the conventional endoscope will be on standby to replace it if necessary, for example in the unlikely event of a failure of the Sirius Robotic Flexible Endoscopic System to work. Your safety is always our priority.

| Risk and complication of the procedure may include, bu | t are not limited to the following |
|---|---|
| <ul> <li>There is no anticipated additional risk for your language.</li> <li>In the unlikely event of an equipment failure conventional endoscope is always on standby to</li> </ul> | of the Sirius Robotic Flexible Endoscopic System, |
| I acknowledge that the above information concerning my discussed with me by the medical staff and I fully understances questions pertinent to my condition and management and staff. | and them. I have been given the opportunity to ask |
| I agree/disagree to participate in this trial. | |
| | Signature: |
| | Date: |